CLINICAL TRIAL: NCT04087538
Title: A Prospective Comparison of Cardiac Troponin T and Troponin I in the Diagnosis of Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Bo Hasselbalch, MD, Herlev Hospital
Other Study IDs: 19000557
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Myocardial Infarction
Keywords: troponin
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated using troponin T
  Interventions: Diagnostic Test: Troponin T and I
- Patients treated using troponin I
  Interventions: Diagnostic Test: Troponin T and I

INTERVENTIONS:
Diagnostic Test: Troponin T and I — Does the use of troponin T or I increase the number of patients referred to coronary angiography

SUMMARY:
The rising number of patients with chest pain without myocardial infarction has made accurate diagnosis important. Unnecessary invasive coronary angiographies are increasingly prevalent. These are both costly and lead to rare but serious adverse events. Recent studies suggest cardiac Troponin I is more cardiac specific than cardiac Troponin T. In this study we will investigate whether using cardiac Troponin I lead to fewer unnecessary procedures in clinical practice (i.e. invasive coronary angiography and non-invasive tests)

ELIGIBILITY:
Inclusion Criteria:

* Admitted to either Herlev-Gentofte or Amager-Hvidovre Hospital
* Clinically suspected of NSTEMI
* Referred to invasive coronary angiography (ICA)
* Recieved at least one measurement of either troponin

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two large acute medical centers will include patients for this study, one that routinely use cTnT (Hvidovre Hospital) and one that routinely uses cTnI (Herlev Hospital).
  Each center will include consecutive patients over a period of 5 months clinically suspected of non-ST segment elevation myocardial infarction (NSTEMI). These patients will undergo serial measurement of either cardiac troponin T (cTnT) or cardiac troponin I (cTnI) as is standard practice. In addition to regular their lab tests, all patients will have extra blood samples set aside for a biobank.
  At the end of the inclusion period, all patients sent to invasive coronary angiography (ICA) will be identified and included in the further analyses. As one center uses cTnT and one uses cTnI, patients will have either biomarker measured upon admission. The other cTn assay will be measured on all samples from the biobank, so every patient has at least one measurement of both cTnT and cTnI.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Specificity for MI | 0
  The difference in specificity of cardiac Troponin and I in detecting patients with significant CAD. The specificity will be defined as the proportion of patients with no significant CAD on ICA correctly identified as low-risk patients and not referred to ICA upon the review by the senior cardiologists
Cost-effectiveness | 0
  The cost-effectiveness of using cardiac Troponin T compared to cardiac Troponin I. This will be defined by the number of patients sent to ICA and the associated costs of this.

SECONDARY OUTCOMES:
Sensitivity for MI | 0
  A safety outcome of difference in sensitivity of cardiac Troponin T and cardiac Troponin I in the detection of patients with significant coronary artery disease. The sensitivity is defined as the proportion of patients with significant coronary artery disease that were referred to ICA upon review by the senior cardiologists
Elevated troponin without CAD | 0
  The difference in the proportion of patients with elevated cardiac Troponin T or cardiac Troponin I above the 99th percentile with no significant CAD on ICA
Number of MIs | 0
  The difference in the number of patients diagnosed with MI for each cardiac Troponin
PPV and NPV | 0
  The difference in positive predictive value and negative predictive value of each cardiac Troponin

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Bispebjerg, Copenhagen
  - Herlev-Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Undecided